CLINICAL TRIAL: NCT04553796
Title: Assessment of Nonalcoholic Fatty Liver Disease in Diabetic and Prediabetic Patients Using Noninvasive Methods.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Melad Fekry Endrawes, principal investigator, Assiut University
Other Study IDs: non alcoholic fatty liver
Record Dates: First submitted 2020-09-12; First posted 2020-09-17 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Non Alcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- diabetic participants: HBA1C : 6.5% or higher Fasting Plasma Glucose : 126 mg/dl or higher Oral Glucose Tolerance Test : 200 mg/dl or higher Random Plasma Glucose Test : greater than or equal to 200 mg/dl
  Interventions: Device: fibroscan
- prediabetic participants: HBA1C : 5.7% to 6.4% Fasting Plasma Glucose : 100 mg/dl to 125 mg/dl Oral Glucose Tolerance Test : 140 mg/dl to 199 mg/dl
  Interventions: Device: fibroscan
- non diabetic participants: HBA1C : less than 5.7% Fasting Plasma Glucose : less than 100 mg/dl Oral Glucose Tolerance Test : less than 140 mg/dl
  Interventions: Device: fibroscan

INTERVENTIONS:
Device: fibroscan — Fibroscan is a non-invasive test that helps assess the health of your liver. Specifically, it uses ultrasound technology to determine the degree of fibrosis or scarring that may be present in your liver from various liver diseases or conditions
  Other Names: Transient Elastography

SUMMARY:
assessment of NAFLD among diabetic, pre-diabetic and non diabetic participants Using Non Invasive Methods.And correlation between lab and radiological methods .

DETAILED DESCRIPTION:
Non alcoholic fatty liver disease (NAFLD) is a major public health problem. with 10-30% prevalence worldwide , and is a common cause of chronic liver disease and the third most common cause of liver transplantation .

NAFLD can range from simple steatosis in the absence of inflammation to nonalcoholic steatohepatitis, liver cirrhosis, and hepatocellular carcinoma (HCC) .

Major risk factors for NAFLD include obesity, hypertension , hyperlipidemia , hypertriglyceridemia , and type-2-diabetes mellitus (T2DM) .

The gold standard in the diagnosis of NAFLD is liver biopsy; however, it is sometimes associated with some complications that include bleeding, bile leak, infection, and other potential life-threatening issues. The accuracy of the MRI, computed tomography, and ultrasound imaging in diagnosis of NAFLD is low; hence, Fibroscan was introduced .

This is a non-invasive, simple-to-perform imaging modality with high accuracy to assess liver stiffness and hepatic fat deposition. Non-invasive diagnosis is based on clinical and biochemical markers, scoring models, and algorithms of methods which have sufficient sensitivity, specificity, and reproducibility .

ELIGIBILITY:
Inclusion Criteria:

* the participants are divided into 3 groups: the diabetic group patients (T2DM) ,the pre-diabetic and the non diabetic one. The diagnosis will be according to the American Diabetes Association (ADA) clinical practice recommendations-2019

Exclusion Criteria:

* patients under the age of 18.
* patients with viral hepatitis (HBV - HCV).
* Subjects with risk of 2nd hepatic steatosis liver disease (excessive alcohol consumption and medications).
* history of liver disease such as (α-1 antitrypsin deficiency, autoimmune hepatitis, drug-induced liver injury, 1ry biliary cirrhosis, 1ry sclerosing cholangitis).
* Body Mass Index (BMI) > 35 (to avoid the possibility of Fibroscan failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants older than 18 years with no definite cause of nafld in our out patient clinic.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
correlation between lab and radiological methods | 2 days
  results of fibroscan, lab investigations include Complete blood picture Fasting plasma glucose (FBG) and Glycated hemoglobin (HbA1C) Liver function tests including ( serum bilirubin , serum albumin , ALT , AST , ALP , prothrombin time and INR ) kidney function tests. Lipid profile including (serum cholesterol and triglycerides ). hepatitis marker (HBs Ag , Anti-HCV Ab). and NAFLD Fibrosis Score will be correlated

CONTACTS AND LOCATIONS:
Overall Officials: lobna a ahmed, professor, Study Chair — Assiut University

REFERENCES:
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Lv S, Jiang S, Liu S, Dong Q, Xin Y, Xuan S. Noninvasive Quantitative Detection Methods of Liver Fat Content in Nonalcoholic Fatty Liver Disease. J Clin Transl Hepatol. 2018 Jun 28;6(2):217-221. doi: 10.14218/JCTH.2018.00021. Epub 2018 Jun 22. PMID 29951367
- [Background] Bazick J, Donithan M, Neuschwander-Tetri BA, Kleiner D, Brunt EM, Wilson L, Doo E, Lavine J, Tonascia J, Loomba R. Clinical Model for NASH and Advanced Fibrosis in Adult Patients With Diabetes and NAFLD: Guidelines for Referral in NAFLD. Diabetes Care. 2015 Jul;38(7):1347-55. doi: 10.2337/dc14-1239. Epub 2015 Apr 17. PMID 25887357
- [Background] Dharmalingam M, Yamasandhi PG. Nonalcoholic Fatty Liver Disease and Type 2 Diabetes Mellitus. Indian J Endocrinol Metab. 2018 May-Jun;22(3):421-428. doi: 10.4103/ijem.IJEM_585_17. PMID 30090738
- [Background] Esterson YB, Grimaldi GM. Radiologic Imaging in Nonalcoholic Fatty Liver Disease and Nonalcoholic Steatohepatitis. Clin Liver Dis. 2018 Feb;22(1):93-108. doi: 10.1016/j.cld.2017.08.005. Epub 2017 Oct 10. PMID 29128063
- [Background] de Ledinghen V, Vergniol J, Foucher J, Merrouche W, le Bail B. Non-invasive diagnosis of liver steatosis using controlled attenuation parameter (CAP) and transient elastography. Liver Int. 2012 Jul;32(6):911-8. doi: 10.1111/j.1478-3231.2012.02820.x. PMID 22672642
- [Background] Castera L, Friedrich-Rust M, Loomba R. Noninvasive Assessment of Liver Disease in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2019 Apr;156(5):1264-1281.e4. doi: 10.1053/j.gastro.2018.12.036. Epub 2019 Jan 18. PMID 30660725
- [Background] Sheth H, Bagasrawala S, Shah M, Ansari R, Olithselvan A, Lakdawala M. The HAALT Non-invasive Scoring System for NAFLD in Obesity. Obes Surg. 2019 Aug;29(8):2562-2570. doi: 10.1007/s11695-019-03880-x. PMID 31016455
- [Background] Wang CC, Jhu JJ. On the Application of Clustering and Classification Techniques to Analyze Metabolic Syndrome Severity Distribution Area and Critical Factors. Int J Environ Res Public Health. 2019 May 6;16(9):1575. doi: 10.3390/ijerph16091575. PMID 31064061
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S13-S28. doi: 10.2337/dc19-S002. PMID 30559228
- [Background] Angulo P, Hui JM, Marchesini G, Bugianesi E, George J, Farrell GC, Enders F, Saksena S, Burt AD, Bida JP, Lindor K, Sanderson SO, Lenzi M, Adams LA, Kench J, Therneau TM, Day CP. The NAFLD fibrosis score: a noninvasive system that identifies liver fibrosis in patients with NAFLD. Hepatology. 2007 Apr;45(4):846-54. doi: 10.1002/hep.21496. PMID 17393509